CLINICAL TRIAL: NCT04515992
Title: Feasibility of Minimal Dose High Intensity Body-weight Circuit Training in Type 2 Diabetics
Brief Title: High Intensity Body-weight Circuit Training in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kennesaw State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: # 18-348
Record Dates: First submitted 2020-08-11; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Body-weight Circuit (HIBC) (Experimental): The at home HIBC intervention program involved the use of both bodyweight and suspension training equipment (TRX® Fit System) with modified movements. The TRX® system was used to modify squats and rows while attached to the top of a door frame.
  Interventions: Behavioral: High Intensity Body-weight Circuit Training (HIBC)

INTERVENTIONS:
Behavioral: High Intensity Body-weight Circuit Training (HIBC) — HIBC Exercise Protocol- The HIBC circuit repetition and order is as follows: modified squats (10 repetitions), modified rows (5 repetitions), crunches (10 repetitions), and modified push-ups (5 repetitions). The exercise sessions involved repeating a series of repetitions of each movement in sequence, and completing as many sequences as possible in good form in the time allotted for the exercise (initially, 5 minutes). Participants were instructed to complete three sessions per week and documented the number of cycles completed. After 3 weeks of consistent training, participants were asked to add a 4th session each week as tolerated. Initially, the HIBC sessions were 5 minutes long, and the duration of the sessions were increased by one minute each week as tolerated beginning in week four, peaking at 10-minutes per session as early as the eighth week of training. Session duration was capped at 10 minutes.

SUMMARY:
Exercise has been shown to be effective at improving fitness, as well as markers of glucose tolerance and control, in persons with type 2 diabetes. Recently, several investigations have demonstrated that improvements are realized by patients with high intensity interval exercise which is characterized by periods of vigorous exercise alternated by periods of moderate exercise. Typical interval training sessions require significantly less time to complete than traditional modes of exercise wherein moderate intensity activity is sustained for some time. This may be especially beneficial to those with type 2 diabetes, as lack of time is a frequently cited reason for not engaging in regular exercise. Bodyweight circuit training carries the potential to similarly improve health and metabolic function in persons with type 2 diabetes, and may do so with even a smaller accumulation of exercise because this type of exercise involves a greater percentage of the trainee's muscle mass compared with common forms of interval training (e.g., treadmill or cycle exercise). The purpose of this study is to quantify the effects of 3-4 sessions per week of bodyweight circuit training sustained for 5-10 minutes per session on health-related physical fitness and glucose tolerance/control in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes of at least 1 year
* hemoglobin A1c level between 6.0% and 10%

Exclusion Criteria:

* Currently engaging in a physical activity
* Currently taking exogenous insulin
* Undertaking a regiment or lifestyle modification intervention.
* Cardiovascular or Pulmonary diseases.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of HbA1c | 16 weeks
  glycosylated hemoglobin, marker of approximate three month blood glucose environment

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kliszczewicz, PhD, Principal Investigator — Kennesaw State University
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Upon publication of research, data will be made publicly available